CLINICAL TRIAL: NCT02572635
Title: A Randomised, Placebo Controlled, Double-blind, Dose Escalation, Single Centre Trial to Evaluate the Safety and Immunogenicity of PnuBioVax Administered on Three Occasions 28 Days Apart at Three Dose Levels in Healthy Adult Subjects.
Brief Title: A Phase I Study to Evaluate the Safety and Immunogenicity of PnuBioVax
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoBiology Limited (Industry)
Collaborators: Simbec Research (Industry); Oxford Therapeutics Consulting Limited (Industry); ORION Clinical Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SPV-001; 2015-002986-51 (EudraCT Number)
Record Dates: First submitted 2015-10-06; First posted 2015-10-09 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Pneumococcal Infection
Keywords: Pneumococcal Infection; Phase I; Immunogenicity; Safety; Vaccination
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 50 µg of PnuBioVax
  Interventions: Biological: PnuBioVax
- Cohort 2 (Experimental): 200 µg of PnuBioVax
  Interventions: Biological: PnuBioVax
- Cohort 3 (Experimental): 500 µg of PnuBioVax
  Interventions: Biological: PnuBioVax
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PnuBioVax — Three administrations (by intramuscular injection) given 28 days apart to 9 subjects.
  Arms: Cohort 1; Cohort 2; Cohort 3
Biological: Placebo — Placebo administered by intramuscular injection to 3 subjects in each cohort. Three administrations given 28 days apart.
  Arms: Placebo

SUMMARY:
Streptococcus pneumoniae is a type of bacteria that can cause infections of the ears, sinuses or lungs. It can also cause more serious infections of the blood or brain. The elderly and young children are more vulnerable to these types of infections.

The vaccines available at present are effective only on a certain number of strains of the bacteria. The PnuBioVax vaccine is being developed to work on a broader range of strains. This study will be looking at the safety and tolerability of the study drug for three different dosages: 50 μg, 200 μg, and 500 μg compared to placebo.

The population eligible to take part in the study are healthy male and female subjects between 18 and 40 years of age.

Volunteers for the study will be recruited through advertisements. Each volunteer will have received an information sheet concerning the study and will have agreed to participate in writing. Volunteers will be given at least 48 hours between reading the information leaflet and agreeing to participate. Only subjects who agree to undertake precautions to avoid pregnancy of either themselves of their partner during the study period will be eligible. Volunteers will give signed consent for their physician to be notified about their participation in the trial.

DETAILED DESCRIPTION:
This is a phase I study to assess the safety and immunogenicity of PnuBioVax administered on three occasions 28 days apart at dose levels of 50 µg, 200 µg, and 500 µg in healthy adult subjects.

The study will involve 8 visits in total; screening period to determine eligibility, 3 treatment periods comprising of an overnight stay at the clinic (days 1, 29 and 57) and 4 outpatient follow up visits (7 days after each dosing period and one on day 85). Volunteers will also be requested to complete a diary card from day 1 to day 85.

36 Volunteers will take part in this study and will be randomly assigned to each sequential dose group as follows:

* Cohort 1: up to 3 doses of 50 µg of PnuBioVax or placebo
* Cohort 2: up to 3 doses of 200 µg of PnuBioVax or placebo
* Cohort 3: up to 3 doses of 500 µg of PnuBioVax or placebo Within each cohort, nine subjects will receive PnuBioVax and three subjects will receive placebo. Each subject will receive administrations of PnuBioVax or placebo on Days 1, 29 and 57.

The lowest dose of PnuBioVax will be evaluated first (i.e. Cohort 1). Dose escalation will only proceed in the subsequent cohorts if blinded safety data (adverse events, injection site reactions, concomitant medication, vital signs and routine laboratory assessments) from day 8 from the 12 subjects in the preceding cohort have been reviewed by the Sponsor and Principal Investigator and are found to be satisfactory. The Sponsor and Principal Investigator will also review the safety data after each subsequent dose to ensure repeat dosing does not give rise to safety issues.

Subjects will be followed up 7 days after each vaccination and also by telephone 14 and 21 days following each vaccination. Subjects will also be requested to record any adverse events in a daily diary. Haematology, biochemistry and vital signs will be measured at each follow up visit (except day 85) and a full safety follow up will be completed 7 days after the third dose (day 64).

Bloods will be drawn for evaluation of the immune response to the PnuBioVax, 28 days following the first, second and third administrations (Days 29, 57 and 85). The blood draw at day 85 will also be used for exploratory analyses.

The presence of autoantibodies will be assessed at screening (baseline level), and day 85 by measurement of anti nuclear antibody (ANA) levels.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female subjects between 18 and 40 years of age (inclusive).
* female subjects of child bearing potential with negative pregnancy test at screening and willing to use 2 effective methods of contraception (i.e. established method of contraception plus condom, or where abstaining from heterosexual intercourse is in line with the preferred and usual lifestyle of the subject) from Day 1 until 3 months after the last dose of PnuBioVax/Placebo.
* male subjects willing to use 2 effective methods of contraception unless anatomically sterile, or where abstaining from heterosexual intercourse is in line with the preferred and usual lifestyle of the subject, from Day 1 until 3 months after the last dose of PnuBioVax/Placebo.
* subjects with a Body Mass Index (BMI) of <30 kg/m2.
* subjects with a negative urinary drugs of abuse screen determined within 28 days of the first dose.
* subjects with negative HIV and Hepatitis B and C results.
* subjects must be willing and able to comply with the requirements of the protocol and must be available to complete the trial, including all follow up visits.
* subject must provide written informed consent to participate in the trial.

Exclusion Criteria:

* any relevant abnormality in medical history examination, vital signs laboratory tests or ECG.
* any reason that would make the assessment of any injection site reaction difficult (e.g. tattoos at injections site, black skin).
* history of migraine or asthma (no inhaler use for 5 years).
* proven diagnosis of pneumonia within last 5 years.
* current smokers.
* history of anaphylaxis or hypersensitivity to previous vaccinations.
* known impairment of the immune system or chronic diseases, e.g. autoimmune diseases, diabetes, cancer.
* anticipation that the subject may require any other vaccination during the trial period.
* subjects who are antinuclear antibody (ANA) positive (above a titre of 1:80).
* subjects with haemoglobin level < 8.4 mmol/ L (males) and <7.8 mmol/L (females).
* palpable cervical or axillary lymph nodes.
* receipt of regular prescribed medication within 28 days of the first trial day and / or receipt of vitamins, minerals, herbal remedies and nutritional supplements within 7 days of the first trial day.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence of all treatment emergent adverse events | Baseline to Day 85
  Number of subjects with adverse events reported from first dosing to last follow up visit.

SECONDARY OUTCOMES:
The proportion of subjects who develop an immune response to PnuBioVax | Baseline to Day 85
  The proportion of subjects with an increase in serum IgG specific for PnuBioVax measured by ELISA on Days 1 (baseline), 29, 57 and 85.

OTHER OUTCOMES:
Measurement of antibody production against specific pneumococcal proteins. | Baseline to Day 85
  Exploratory analyses measuring change from baseline in serum IgG against nine pneumococcal antigens by electrochemiluminescence detection in an immunoassay.
Measurement of the percentage inhibition by serum of the haemolytic activity of pneumolysin. | Baseline to Day 85
  Exploratory assay to determine the ability of antibodies in serum to neutralise the haemolytic activity of pneumolysin.
Measurement of IL-17 production following stimulation of peripheral blood mononuclear cells with PnuBioVax. | Baseline to Day 85
  Exploratory analysis to measure the ability of peripheral blood mononuclear cells to produce IL-17 following stimulation with PnuBioVax measured by ELISA and ELISPOT.
Measurement of the opsonophaocytic activity of serum antibodies against a target panel of S. pneumoniae strains | Baseline to Day 85
  Exploratory analysis measuring change from baseline in the percentage killing of multiple strains of S. pneumoniae using opsonophagocytic activity assays.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bailey, Bsc, PhD, Study Director — Sponsor (ImmunoBiology Ltd)
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, Glamorgan, United Kingdom

REFERENCES:
- [Derived] Entwisle C, Hill S, Pang Y, Joachim M, McIlgorm A, Colaco C, Goldblatt D, De Gorguette D'Argoeuves P, Bailey C. Safety and immunogenicity of a novel multiple antigen pneumococcal vaccine in adults: A Phase 1 randomised clinical trial. Vaccine. 2017 Dec 18;35(51):7181-7186. doi: 10.1016/j.vaccine.2017.10.076. Epub 2017 Nov 10. PMID 29132988